CLINICAL TRIAL: NCT03808194
Title: The Lotto to Link Study: A Prospective, Interventional, Randomized Study of Conditional Incentives to Engage HIV-positive Men in HIV Care in KwaZulu-Natal, South Africa
Brief Title: Lotto to Link Study: A Prospective, Interventional, Randomized Study of Conditional Incentives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ruanne Barnabas, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STUDY00000036; 5R21MH110026 (NIH)
Record Dates: First submitted 2019-01-03; First posted 2019-01-17 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Incentives; HIV Infections; ART
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: HIV-positive men who meet the study eligibility criteria will be randomized to one of two study arms: 1) Optimized ART linkage package, or 2) Optimized ART linkage package + conditional lottery incentive.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimized ART linkage package (Active Comparator): Participants in this arm will receive a clinic referral card and text messages to support linkage to ART.
  Interventions: Other: Optimized ART linkage package
- Conditional lottery incentive (Experimental): Participants in this arm will receive a clinic referral card and text messages to support linkage to ART and will be entered into a lottery each time they meet the following conditions: visited the clinic by month 1, initiated treatment by month 3, and achieved viral suppression by month 6
  Interventions: Other: Conditional lottery incentive

INTERVENTIONS:
Other: Conditional lottery incentive — Participants in the lottery incentive arm must fulfill the following criteria to be entered into the lottery. Participants must visit the clinic by month 1, initiate ART by month 3 and achieve viral suppression by month 6. Participants in this arm will be eligible to win the lottery.
  Arms: Conditional lottery incentive
Other: Optimized ART linkage package — Optimized ART linkage package
  Arms: Optimized ART linkage package

SUMMARY:
In this study the investigators will adapt and strengthen, test effectiveness, and explore implementation of conditional lottery incentive linkage strategies to engage men in HIV care and ART in KwaZulu-Natal, South Africa.

DETAILED DESCRIPTION:
Of the 2.6 million South Africans on antiretroviral therapy (ART)1 only a third are men, despite men making up 45% of HIV-positive persons.2 HIV-positive men are underrepresented throughout the HIV prevention and care continuum, being less likely to test, link to care, initiate ART, and more likely to be lost to follow-up. Few strategies have focused on men, and when they have they have not been successful. Even with community-based HIV testing, referral, text message reminders, and lay-counselor support (an optimized testing and linkage to care package), doctors are only able to achieve 60% linkage to HIV care and ART among men. HIV-positive men who are not in care are at risk for HIV-associated morbidity and mortality, and their HIV-negative partners are at risk of HIV acquisition. Innovative strategies are needed to motivate HIV-positive men to engage in care, and specifically to initiate and adhere to ART.

Introducing a gamble, the chance of winning a lottery, into linkage to HIV care interventions could make engagement in care more attractive to men. Men are often risk-takers and linking to care successfully is a gamble: start ART vs. risk no ART. A lottery incentive strategy has been successfully used to increase uptake of HIV prevention; in one recent example, lottery incentives, conditioned on being STI (sexually transmitted infection) negative, decreased HIV incidence by 60% among 'risk-loving' individuals in Lesotho, demonstrating one of the largest effects to date of a behavioral intervention for HIV prevention. Given this prevention success, the investigators hypothesize that lottery incentives have the potential to overcome both structural and behavioral factors for linking HIV positive men to care, addressing logistical challenges and risk preferences specific to men. For scale-up and implementation, the investigators need to sculpt the content of lottery incentive strategies as well as the approach to identify men not in care for whom lottery incentives are likely to work.

In this study the investigators will adapt and strengthen, test effectiveness, and explore implementation of conditional lottery incentive linkage strategies to engage men in HIV care and ART in KwaZulu-Natal, South Africa (the Lotto to Link Study). With the investigators experienced, multi-disciplinary team, the investigators have drawn on their previous successful community-based counseling and testing and linkage to prevention and care work to strengthen linkage strategies for HIV-positive ART eligible men who are not in care.

The investigators will do 1) qualitative interviews to inform the study design, 2) conduct an individual randomized study of conditional lottery incentives compared to an optimized linkage package for HIV-positive men, and 3) finally, estimate the costs associated with conditional incentives and retention in care.

ELIGIBILITY:
Inclusion Criteria:

* Reside in the study community for the duration of follow-up
* Must be 18 years or older
* Able and willing to provide informed consent for study procedures
* HIV-positive men must be eligible for ART by national guidelines and not on ART
* Access to confidential text messaging

Exclusion Criteria:

• There are no separate exclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Number of men virally suppressed after 6 months | 6 months
  Conditional lottery incentives, above and beyond an optimized linkage package, will increase the uptake of clinic visits, ART initiation, and viral suppression among HIV-positive men not yet in care.

SECONDARY OUTCOMES:
Number of men who have a positive alcohol or drug test | 6 months
  Men who currently use drugs, consume more than the recommended amount of alcohol on an ongoing basis, or report depression and anxiety are less likely to link to care, stay retained in care, and achieve virologic suppression.

CONTACTS AND LOCATIONS:
Overall Officials: Ruanne V Barnabas, MD, Principal Investigator — University of Washington
Locations (1):
- HSRC Sweetwaters, Sweetwaters, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barnabas RV, van Heerden A, McConnell M, Szpiro AA, Krows ML, Schaafsma TT, Ngubane T, Nxele RB, Joseph P, Baeten JM, Celum CL, van Rooyen H. Lottery incentives have short-term impact on ART initiation among men: results from a randomized pilot study. J Int AIDS Soc. 2020 Jun;23 Suppl 2(Suppl 2):e25519. doi: 10.1002/jia2.25519. PMID 32589342